CLINICAL TRIAL: NCT07355218
Title: A Phase 3, Randomized, Double-Blind,Placebo-Controlled Parallel Study to Evaluate the Efficacy and Safety of Enpatoran in Participants With Active Cutaneous Manifestations of Lupus Erythematosus With or Without Systemic Disease Receiving Standard of Care (ELOWEN-2)
Brief Title: A Study of Enpatoran in Participants With Cutaneous Manifestations of Lupus With or Without Systemic Disease (ELOWEN-2)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS504908_0008; 2025-524855-30-00 (EU CTIS Number); 169831 (Other: IND)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Systematic Lupus Erythematosus; Cutaneous Lupus Erythematosus
Keywords: Toll-like Receptor 7; Toll-like Receptor 8; Adults; SLE; CLE; Lupus; Discoid lupus erythematosus; Subacute cutaneous lupus erythematosus; M5049; Enpatoran; Cutaneous manifestations; Lupus erythematosus; Acute cutaneous lupus erythematosus; Systemic lupus erythematosus; Interferon gene signature
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enpatoran (Experimental)
  Interventions: Drug: Enpatoran; Drug: Standard of care (SoC)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Standard of care (SoC)

INTERVENTIONS:
Drug: Enpatoran — Participants will receive a dose of Enpatoran orally twice daily from Day 1 to Day 168.
  Other Names: M5049
  Arms: Enpatoran
Drug: Placebo — Participants will receive a single oral dose of a placebo matching Enpatoran tablet twice daily from Day 1 to Day 168.
  Arms: Placebo
Drug: Standard of care (SoC) — Participants will receive Investigator-recommended SoC.

SUMMARY:
The purpose of this global, multicenter, Phase 3 study is to evaluate the efficacy and safety of enpatoran over 24 weeks in participants with active cutaneous manifestations of lupus erythematosus with or without systemic disease. Study details include:

Study Duration: Up to 35 weeks. Treatment Duration: 24 weeks. Visit Frequency: every 4 weeks, with the exception of the Week 2 televisit. Study Intervention Name: Enpatoran, Placebo.

Intervention Form: Film-coated tablet.

ELIGIBILITY:
Inclusion Criteria

* Vaccinations are up to date according to local guidelines/recommendations. Recombinant zoster vaccination is encouraged but not mandatory.
* Participants with diagnosis of Discoid Lupus Erythematosus (DLE) and/or Subacute Cutaneous Lupus Erythematosus (SCLE) documented in medical history, with or without Systemic Lupus Erythematosus (SLE).
* Participants with active Acute Cutaneous Lupus Erythematosus (ACLE) as sole cutaneous manifestations is allowed in the presence of SLE and should be present for at least 6 weeks prior to the Screening visit.
* Participants with diagnosis of SLE fulfilling the European Alliance of Associations for Rheumatology (EULAR)/American College of Rheumatology (ACR) 2019 classification criteria, must have active DLE and/or SCLE and/or ACLE.

For participants with SLE:

* Participants with diagnosis of SLE and fulfill EULAR/ACR 2019 classification criteria.
* Participants with disease duration (cutaneous disease and, where applicable, SLE) of >= 6 months from time of diagnosis to Screening.
* Participants with CLASI-A score >= 8 at Screening and Day 1 visits.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria

* Participants with primary diagnosis of autoimmune rheumatic disease (e.g., systemic sclerosis, rheumatoid arthritis) other than Cutaneous Lupus Erythematosus (CLE) and SLE.
* Participants with any condition including dermatological diseases other than cutaneous manifestations of lupus (e.g. psoriasis), any uncontrolled disease (e.g. asthma, chronic obstructive pulmonary disease, interstitial lung disease, bronchiectasis, pulmonary arterial hypertension), or life-threatening manifestations of lupus (e.g. active systemic vasculitis) that in Investigator's or Sponsor/designee's opinion constitutes inappropriate risk or contraindication for participation.
* Participants with drug-induced lupus (SLE or CLE).
* Participants with active lupus nephritis on induction therapy, or induction therapy completed within 3 months of the Screening visit (stable maintenance therapy with either mycophenolate azathioprine or an oral calcineurin inhibitor is allowed).
* Participants with Urine Protein-to-Creatinine Ratio (UPCR) greater than (>) 339 milligrams per millimole (mg/mmol), and/or estimated Glomerular Filtration Rate (eGFR) less than 40 milliliters per minute per 1.73 square meters of body surface area (mL/min/1.73 m^2), as calculated by the Modification of Diet in Renal Disease (MDRD) equation.
* Participants with any active signs, symptoms, or diagnoses considered related to Central Nervous System (CNS) lupus within the past 3 months, or any history of uncontrolled seizures.
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2029-03-19 (Estimated); Study Completion 2029-03-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) 70 Response, Defined as >= 70 Percent (%) Decrease in CLASI-A Score From Baseline | At Week 24

SECONDARY OUTCOMES:
Percentage of Participants With British Isles Lupus Assessment Group Based Composite Lupus Assessment (BICLA) Response | At Week 24
  A BICLA response is defined as British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004) -improvement without worsening (A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and less than or equal to [<=] 1 new B.); Here, score A ("Active"): Severely active disease; score B ("Beware"): Moderately active disease; score C ("Contentment"): Mild stable disease; score D ("Discount"): Inactive now but previously active; -no worsening in disease activity (no new BILAG 2004 A scores and <= 1 new B score); -no worsening of total Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score from Baseline; -no significant deterioration (less than [<] 10% worsening) in visual analog Physician's Global Assessment (PGA) and -no treatment failure i.e. protocol-prohibited medications as determined by Endpoint Adjudication Committee (EAC) or premature discontinuation from study treatment).
Number of Participants With Treatment Emergent adverse events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESI) | From Day 1 to Week 24
Number of Participants With Abnormal (greater than and equal to [>=] Grade 3) laboratory parameters | From Day 1 to Week 24
Percentage of Participants With CLASI-A less than and equal to (<=) 3 at Week 24 | At Week 24
  CLASI-A assesses the signs of CLE disease activity including erythema, scale, and hypertrophy, active alopecia, and mucous membrane disease, Scores range from 0 to 70 points for CLASI-A score. Mild, moderate, and severe disease corresponds with CLASI activity score ranges of 0 to 9, 10 to 20, and 21 to 70, respectively. Higher scores indicate more disease activity.
Percentage of Participants With CLASI-50 Response, Defined as >=50% Decrease in CLASI-A Score From Baseline | At Weeks 4 and 24
Percentage of Participants With Clinically Meaningful Corticosteroid (CS) Reduction | Day 1 up to Week 12 and thereafter upto Week 24
  Clinically meaningful CS reduction, is defined as reduction of daily prednisone-equivalent dose from >= 10 milligrams (mg) at Day 1 to <= 5 mg by the Week 12 visit and sustained through Week 24.
Change from Baseline in Worst Itch Numeric Rating Scale (NRS) Score at Week 24 | Baseline and at Week 24
  The Worst Itch NRS is a self-rated single item scale designed for assessing worst itch in the past 7 days. The scale utilizes 11-point NRS, scored from of 0 (no itch) to 10 (worst imaginable itch).
Change from Baseline in CLASI-A Erythema at Week 24 | Baseline and at Week 24
  CLASI-A assesses the signs of CLE disease activity including erythema, scale, and hypertrophy, active alopecia, and mucous membrane disease, Scores range from 0 to 70 points for CLASI-A score. Mild, moderate, and severe disease corresponds with CLASI activity score ranges of 0 to 9, 10 to 20, and 21 to 70, respectively. Higher scores indicate more disease activity.
Change from Baseline in CLASI-A Scale/Hypertrophy at Week 24 | Baseline and at Week 24
  CLASI-A assesses the signs of CLE disease activity including erythema, scale, and hypertrophy, active alopecia, and mucous membrane disease, Scores range from 0 to 70 points for CLASI-A score. Mild, moderate, and severe disease corresponds with CLASI activity score ranges of 0 to 9, 10 to 20, and 21 to 70, respectively. Higher scores indicate more disease activity.
Change from Baseline in CLASI-A Alopecia at Week 24 | Baseline and at Week 24
  CLASI-A assesses the signs of CLE disease activity including erythema, scale, and hypertrophy, active alopecia, and mucous membrane disease, Scores range from 0 to 70 points for CLASI-A score. Mild, moderate, and severe disease corresponds with CLASI activity score ranges of 0 to 9, 10 to 20, and 21 to 70, respectively. Higher scores indicate more disease activity.
Percentage of Participants With a Cutaneous Lupus Activity Investigator's Global Assessment-Revised (CLA-IGA-R OMC) Score of 0 or 1 and at Least a 1-Point Reduction at Week 24 | At Week 24
  The CLA-IGA-R is assessed by the investigator, who assigns rater to assign scores to 3 individual domains (e.g. erythema, other morphologic characteristics - OMC [scales, edema)/infiltration and secondary change (vesicles, erosion, crusting)] and follicular activity). Clinicians assess the severity of the first 2 domains of erythema and OMC from 0 (Clear) to 4 (Severe); they assess the severity of the third domain of follicular activity as "absent" or "present." Higher scores indicate more disease activity.
Percentage of Participants with BILAG Moderate to Severe Flares | up to Week 24
Time to First Moderate/Severe BILAG Flare | Day 1 through Week 24
  Median time to first moderate or severe BILAG Flare will be calculated.
Percentage of Participants with Corticosteroid (CS) reduction of Daily Prednisone Equivalent Dose | Day 1 up to 24 weeks
  CS reduction is defined as of daily prednisone-equivalent dose from >= 10 milligrams per day (mg/day) at Day 1 to <= 5 mg/day and sustained for 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Research Site, Darmstadt, Germany

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union.
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html